CLINICAL TRIAL: NCT03016923
Title: An Evaluation of the Effectiveness of Functional Electrical Stimulation Paired With Intensive Therapy to Improve Hand Function in Children With Hemiplegic Cerebral Palsy
Brief Title: Functional Electrical Stimulation (FES) for Upper Extremity Hemiplegia in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-549
Record Dates: First submitted 2016-04-25; First posted 2017-01-11 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2016-04

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; hemiplegia; fes; grasping
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FES Therapy (Experimental): FES therapy will be administered over the course of 1 hour sessions that will be take place 3 times per week over 16 weeks, for a total of 48 sessions.
  Interventions: Device: FES Therapy

INTERVENTIONS:
Device: FES Therapy — FES therapy will be administered over the course of 1 hour sessions that will be take place 3 times per week over 16 weeks, for a total of 48 sessions.

SUMMARY:
The proposed pilot study seeks to explore the effectiveness of Functional Electrical Stimulation (FES) to improve upper limb function in children and youth (aged 6 to 18 years) with hemiplegic cerebral palsy, as measured by the QUEST grasp score and other secondary outcome measures obtained pre- and post-intervention in a case series study design.

DETAILED DESCRIPTION:
Functional electrical stimulation (FES) has increasingly gained interest as a therapeutic intervention for the improvement of motor function in individuals with disabilities. FES involves the administration of electrical pulses to stimulate motor neurons and initiate muscle contractions, It has been used primarily for individuals with spinal cord injury or those who have experienced a stroke leading to the loss of or decreased motor function of the limbs. The repeated application of FES to the affected limb has been shown to enable individuals with hemiplegia to voluntarily control movements of the affected upper limb. A new FES system, has recently been developed and indicated for use for the improvement of arm and hand function in patients with hemiplegia due to stroke or spinal cord injury. FES is a non-invasive therapy that involves transcutaneous delivery of electrical stimulation to the affected upper limb, patient participation and the assistance of therapists to improve voluntary arm and hand movements such as reaching and grasping.

The new FES system has shown effectiveness in both adults with acute stroke and children with chronic acquired stroke. In a randomized controlled trial, FES paired with intensive therapy compared to intensive therapy alone was shown to significantly improve hand function for adults with acute stroke. Participants in the trial had limited mobility or complete immobility of the affected arm and those who received FES paired with intensive therapy had clinically significant improvements in hand movements compared to those who only received intensive therapy. Recently, transcutaneous FES paired with intensive hand therapy (3 one-hour sessions per week for 16 weeks) has more recently been shown to improve hand function in children with chronic acquired stroke.

The efficacy of FES seen in patients with stroke opens up the possibility for its use in other similar populations, including children with hemiplegic cerebral palsy (HCP). However, there is currently limited research on the efficacy of FES with this population. In a preliminary study, the use of FES alone over a treatment period of 6 weeks in children with HCP was shown to significantly improve wrist movement. However, most of the research to date on the effects of FES on children with HCP has been focused on gait and lower limb function. There is currently a lack of evidence on the effectiveness of FES paired with intensive therapy on hand function in children with HCP. FES paired with intensive therapy holds significant potential to improve the hand function of children with HCP and warrants further investigation.

Therefore, the proposed research seeks to address two main objectives:

1. To investigate the effectiveness of FES to improve upper limb function in children with HCP.
2. To assess the effects of FES on upper limb function in children with HCP at six months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hemiplegic CP
* Age between 6 to 18 years
* Ability to cooperate, understand and follow instructions during the administration of FES paired with intensive hand therapy
* Baseline total QUEST score between 20-80 out of 100 points
* Be seizure-free for a required period of at least 1 year with or without medication , and have no prior history of known cardiac arrhythmias/stimulants
* No pacemaker or implanted metallic or electronic device
* No edema, skin rash, allergy or wound on the affected upper limb where FES will be administered.
* No Botulinum toxin upper limb injections within 6-months of study entry, and no Constraint-induced movement therapy (CIMT) within 4 months of study entry. Participants should also refrain from receiving these treatments throughout the duration of the study.

Exclusion Criteria:

* The participant's forearm is too small to accommodate the standard FES electrodes.
* The participant's muscles do not respond to the electrical stimulation as tested at the baseline assessment visit. Response to electrical stimulation will be tested at the baseline visit and is described in detail in the section entitled "Muscle Responsiveness Testing" below. Based on the Muscle Responsiveness Testing procedures and criteria, the withdrawal criteria for non-response to electrical stimulation is defined as:

  1. More than 3 muscle groups out of 11 not- responding to FES or
  2. The participant reports a discomfort level score of 8 or 10 on the FACES scale (Appendix A) for any of the 11 muscle groups.
* Participant receives any other active occupational therapy or hemiplegic hand intervention during the FES intervention period.
* Participant attends less than 36/48 FES intervention sessions.
* Participant develops new-onset seizures during the FES intervention period.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2016-03; Primary Completion 2017-08-25 (Actual); Study Completion 2017-08-25 (Actual)

PRIMARY OUTCOMES:
Quality of Upper Extremities Skills Test (QUEST) as a measure of Movement patterns and hand function | Change from Baseline (i.e, prior to intervention), at 4 months post-intervention, and at 6 months post-intervention

SECONDARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) as a measure of change in a child's self-perception of occupational performance over time | Change from Baseline (i.e, prior to intervention), at 4 months post-intervention, and at 6 months post-intervention
Grip Strength Test as a measure of hand and forearm muscular strength | Change from Baseline (i.e, prior to intervention), at 4 months post-intervention, and at 6 months post-intervention
Jebsen-Taylor Test of Hand Function (JTTHF) as a measure of hand functions required in activities of daily living | Change from Baseline (i.e., prior to intervention), at 4 months post-intervention, and at 6 months post-intervention. JTTHF will also be assessed at 4 weeks, 8 weeks, 12 weeks, and 16 weeks during the intervention period.
Children's Hand-use Experience Questionnaire (CHEQ) as a measure of children's experience in using the affected hand in bi-manual activities | Change from Baseline (i.e, prior to intervention), at 4 months post-intervention, and at 6 months post-intervention
Proprioception Task as a measure of joint-position sense | Change from Baseline (i.e, prior to intervention), at 4 months post-intervention, and at 6 months post-intervention
Two-point Orientation Discrimination (2POD) as a measure of tactile spatial acuity | Change from Baseline (i.e, prior to intervention), at 4 months post-intervention, and at 6 months post-intervention
Stereognosis Test as a measure of is the ability to recognize and identify common objects through tactile manipulation without the use of visual cues | Change from Baseline (i.e, prior to intervention), at 4 months post-intervention, and at 6 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Darcy Fehlings, MD, MSc, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kapadia NM, Nagai MK, Zivanovic V, Bernstein J, Woodhouse J, Rumney P, Popovic MR. Functional electrical stimulation therapy for recovery of reaching and grasping in severe chronic pediatric stroke patients. J Child Neurol. 2014 Apr;29(4):493-9. doi: 10.1177/0883073813484088. Epub 2013 Apr 12. PMID 23584687
- [Background] Thrasher TA, Zivanovic V, McIlroy W, Popovic MR. Rehabilitation of reaching and grasping function in severe hemiplegic patients using functional electrical stimulation therapy. Neurorehabil Neural Repair. 2008 Nov-Dec;22(6):706-14. doi: 10.1177/1545968308317436. PMID 18971385
- [Background] Kawashima N, Popovic MR, Zivanovic V. Effect of intensive functional electrical stimulation therapy on upper-limb motor recovery after stroke: case study of a patient with chronic stroke. Physiother Can. 2013 Winter;65(1):20-8. doi: 10.3138/ptc.2011-36. PMID 24381377
- [Background] Sheffler LR, Chae J. Neuromuscular electrical stimulation in neurorehabilitation. Muscle Nerve. 2007 May;35(5):562-90. doi: 10.1002/mus.20758. PMID 17299744
- [Background] Quandt F, Hummel FC. The influence of functional electrical stimulation on hand motor recovery in stroke patients: a review. Exp Transl Stroke Med. 2014 Aug 21;6:9. doi: 10.1186/2040-7378-6-9. eCollection 2014. PMID 25276333
- [Background] Meadmore KL, Exell TA, Hallewell E, Hughes AM, Freeman CT, Kutlu M, Benson V, Rogers E, Burridge JH. The application of precisely controlled functional electrical stimulation to the shoulder, elbow and wrist for upper limb stroke rehabilitation: a feasibility study. J Neuroeng Rehabil. 2014 Jun 30;11:105. doi: 10.1186/1743-0003-11-105. PMID 24981060
- [Background] Golomb MR, Garg BP, Saha C, Azzouz F, Williams LS. Cerebral palsy after perinatal arterial ischemic stroke. J Child Neurol. 2008 Mar;23(3):279-86. doi: 10.1177/0883073807309246. PMID 18305317
- [Background] Prosser LA, Curatalo LA, Alter KE, Damiano DL. Acceptability and potential effectiveness of a foot drop stimulator in children and adolescents with cerebral palsy. Dev Med Child Neurol. 2012 Nov;54(11):1044-9. doi: 10.1111/j.1469-8749.2012.04401.x. Epub 2012 Aug 27. PMID 22924431
- [Background] Wright PA, Granat MH. Therapeutic effects of functional electrical stimulation of the upper limb of eight children with cerebral palsy. Dev Med Child Neurol. 2000 Nov;42(11):724-7. doi: 10.1017/s0012162200001341. PMID 11104342
- [Background] Postans NJ, Granat MH. Effect of functional electrical stimulation, applied during walking, on gait in spastic cerebral palsy. Dev Med Child Neurol. 2005 Jan;47(1):46-52. doi: 10.1017/s0012162205000083. PMID 15686289
- [Background] Staudt M, Gerloff C, Grodd W, Holthausen H, Niemann G, Krageloh-Mann I. Reorganization in congenital hemiparesis acquired at different gestational ages. Ann Neurol. 2004 Dec;56(6):854-63. doi: 10.1002/ana.20297. PMID 15562409